CLINICAL TRIAL: NCT02612948
Title: Quetiapine for Delirium Prophylaxis in High-risk Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Brian Daley, Professor, University of Tennessee Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3709
Record Dates: First submitted 2015-11-19; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Psychomotor Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Standard care for delerium
- Quetiapine (Active Comparator): Quetiapine therapy was initiated at 12.5 mg twice daily a. After thefirst dose of quetiapine 12.5 mg, the regimen could then be adjusted by the rounding surgeon. If the surgeon felt benefit from receiving a higher dose of quetiapine the dose could then be increased. Quetiapine was discontinued if adverse events (torsades de pointes or other ventricular tachycardias) occurred. All patients receiving at least one dose of quetiapine were included in the final intention-to-treat analyses. All prescribing decisions were left to the discretion of the rounding surgeon and were not mandated as part of the study.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — escalating dose to prevent delerium.
  Other Names: Seroquel
  Arms: Quetiapine

SUMMARY:
Scheduled, low-dose quetiapine is effective in preventing delirium in high-risk critically ill, trauma/surgical patients. Prophylaxis also reduced ventilator duration and ICU length of stay.

DETAILED DESCRIPTION:
Objective: To evaluate the efficacy of scheduled quetiapine for delirium prophylaxis in critically ill, trauma/surgical patients identified as high-risk for delirium utilizing a validated prediction model.

Design: Prospective, open-label, single-center study. Setting: Trauma/surgical intensive care unit at an academic medical center. Patients: Eighty two adult trauma/surgical patients who were admitted to the intensive care unit and were at high-risk for the development of delirium (PRE-DELIRIC Score ≥50%, past medical history of dementia, past medical history of alcohol misuse, or past medical history of drug abuse).

Interventions: Patients were randomized by unit location to receive pharmacologic prophylaxis for delirium (quetiapine 12.5 mg every 12 hours) or no pharmacologic prophylaxis for delirium within forty-eight hours of admission to the intensive care unit.

Measurements: The primary end point was the incidence of delirium during admission to the intensive care unit (ICU). Secondary end points included time to onset of delirium, ICU and hospital lengths of stay, ICU and hospital mortality, duration of mechanical ventilation, and adverse events. Delirium was assessed using the confusion assessment method for the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Trauma/surgical patients admitted to the trauma/surgical ICU

Exclusion Criteria:

* sustained RASS of -4/-5 during the complete ICU admission
* presence of a condition preventing delirium assessment
* anticipated or known ICU length of stay of less than 48 hours
* taking antipsychotics prior to admission
* history of schizophrenia, epilepsy, parkinsonism, or levodopa treatment
* primary neurologic event/injury with GCS ≤ 9 during the first 48 hours of ICU
* current treatment with a continuous infusion neuromuscular blocking agent
* pregnancy
* screened positive for delirium upon admission to the ICU.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of delerium | One year
  ICU length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Brian Daley, Principal Investigator — University General Surgeons, P.C.
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States